CLINICAL TRIAL: NCT05287516
Title: Use of a Digital Visual Analog Scale With Smart Phones for Appetite Measures in the Real World: A Validation Study
Brief Title: Validation of a Digital Visual Analogue Scale for Appetite Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Mills (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2022/03/11
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Healthy
MeSH Terms: interventions — Breakfast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breakfast meal with 460 kcal (Experimental)
  Interventions: Other: Breakfast meal
- Breakfast meal with 230 kcal (Active Comparator)
  Interventions: Other: Breakfast meal

INTERVENTIONS:
Other: Breakfast meal — A meal consisting of breakfast biscuits and water.

SUMMARY:
The objective of the study is to validate a newly developed digital visual analog scales with a mobile app for measuring human appetite and compare it with a traditional paper-based visual analog scales for appetite measurement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-70 years.
* Body mass index 20-29.9 kg/m² (based on self-reported weight and height).
* Understand the study procedures.
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial.
* Willing to follow study procedures on test days.
* Willing to abstain from strenuous exercise, consuming alcoholic drinks 24 hours before the test day.
* Willing to provide informed consent to participate in the study.

Exclusion Criteria:

* Pregnant or lactating women, or women who are planning to become pregnant during the study
* Known food allergies, sensitivity, or intolerance to any food or food ingredients
* Participating in another clinical trial for food, investigational drug, nutritional supplement, or lifestyle modification
* Taking medications that affect appetite, metabolism, or blood pressure
* Presence of acute diseases or infection
* Presence or history of chronic diseases
* Diagnosed with eating disorders
* Restraint eaters
* Lost or gained 5 pounds or more in the past 3 months
* On a weight-loss diet, or undergoing intermittent fasting
* COVID-19 infection in the past 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve for Hunger 0-240 min | 0-240 min
  Area Under the Curve for Hunger 0-240 min
Area Under the Curve for Fullness 0-240 min | 0-240 min
  Area Under the Curve for Fullness 0-240 min
Area Under the Curve for Desire to Eat 0-240 min | 0-240 min
  Area Under the Curve for Desire to Eat 0-240 min
Area Under the Curve for Prospective Consumption 0-240 min | 0-240 min
  Area Under the Curve for Prospective Consumption 0-240 min
Area Under the Curve for Satiety 0-240 min | 0-240 min
  Area Under the Curve for Satiety 0-240 min

CONTACTS AND LOCATIONS:
Locations (1):
- Remote study, No physical facility, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No